CLINICAL TRIAL: NCT05297864
Title: Phase II Trial of Niraparib in Patients With Recurrent Glioma
Brief Title: PARP Inhibition for Gliomas (PI-4G or π4g)
Acronym: OU-SCC-PI-4G
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder terminated funding.
Sponsor: University of Oklahoma (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-PI-4G
Record Dates: First submitted 2022-03-09; First posted 2022-03-28 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Glioblastoma; Recurrent Astrocytoma; Recurrent Oligodendroglioma; Recurrent Glioma
Keywords: high grade gliomas
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Niraparib Treatment (Experimental): Patients will be treated with individualized starting dose of Niraparib.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — The starting dose will be 300 mg niraparib (or modified according patient weight and platelet count), taken orally once a day for each cycle of 28 days.

SUMMARY:
The purpose of this study is to determine what effects (good and bad) niraparib has on patients with recurrent brain cancer.

DETAILED DESCRIPTION:
Patients will have tests and exams to see if they are eligible for the clinical trial. If found eligible, the patient will receive treatment with niraparib in the form of capsules taken every day for the first 28 days. If this dose is tolerated well, the patients will continue to take the capsules and more patients will be enrolled on the study.

Patients will continue treatment with niraparib while on the study unless there is evidence of tumor growth or they experience unacceptable side effects.

Patients will be monitored during treatment with tests and exams and after treatment completion for up to four years from the time they enrolled on the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand and willing to sign the informed consent form.
2. Patients must be ≥ 18 years of age.
3. Patients must have histologically proven high-grade gliomas - GBM, Astrocytoma, or Oligodendroglioma (glioma WHO Grade III or IV) that is now recurrent by MRI or surgical pathology.
4. Patients must have measurable or evaluable lesions by RANO.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Patient has archival tumor tissue available; or a fresh biopsy of recurrent or persistent tumor must be obtained for molecular assay by myChoice test (Myriad Genetics) prior to study treatment initiation. Patient will be requested to share reports from any prior genetic testing with the study investigators.
7. Participants have systolic BP< 140 mmHg or diastolic BP <90 mmHg that has been adequately treated or controlled.
8. Have adequate organ function defined per protocol.
9. Be able to take oral medications
10. Life expectancy ≥ 3 months, allowing adequate follow up of toxicity evaluation and antitumor activity.
11. Female patient, if of childbearing potential, has a negative serum pregnancy test within 72 hours of taking study medication and agrees to abstain from activities that could result in pregnancy from enrollment through 180 days after the last dose of study treatment or is of nonchildbearing potential.
12. Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient. In addition, men must not donate sperm during niraparib therapy and for 90 days after receiving the last dose of niraparib.
13. Patient must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.
14. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
15. Participant receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy.

Exclusion Criteria:

1. Patient has a known additional malignancy that progressed or required active treatment within the last 3 years (exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer).
2. Prior treatment with a known poly (ADP-ribose) polymerase (PARP) inhibitor
3. Participants with human immunodeficiency virus (HIV) with detectable viral load. Participants with HIV on effective anti-retroviral therapy with documented undetectable viral load and CD4 count ≥ 350 within 6 months of the first dose of study treatment are eligible for this trial.
4. Known active hepatitis B or hepatitis C.
5. Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
6. Participant is pregnant or expecting to conceive while receiving study treatment and/or for up to 180 days after the last dose of study treatment. Patient currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first dose of study drug.
7. Received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 4 weeks
8. Patients must not have a known hypersensitivity to the components of niraparib or the excipients (lactose monohydrate and magnesium stearate).
9. Patients must not have had major surgery within 4 weeks (including craniotomy) of starting the study and patient must have recovered from any effects of any major surgery. Stereotactic biopsy by burr hole is considered a minor surgery, and those patients undergoing this surgery will be eligible for the study 2 weeks post-procedure.
10. Patients must not have had radiotherapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
11. Patients must not have received a transfusion (platelets or red blood cells), colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) ≤ 4 weeks of the first dose of study treatment.
12. Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
13. Participants have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
14. Participants have received live vaccine within 30 days of planned start of study randomization.
15. Patients have medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
16. Any medical condition not yet specified above that is considered to possibly, probably or definitely interfere with study procedures, including adequate follow-up and compliance and/or would jeopardize safe treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Battiste, MD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multisite study, but only enrolled participants at University of Oklahoma Health Sciences Center Stephenson Cancer Center (OUHSC SCC). The study activated at SCC on 4/14/2022 and the last patient went off study on 2/6/2024. The first patient enrolled on 6/9/2022 and the last patient enrolled on 9/28/2023.
Pre-assignment Details: Of the 15 enrolled participants, 9 met inclusion criteria and were evaluable.
Groups:
- Niraparib Treatment: Patients will be treated with individualized starting dose of Niraparib.
  Niraparib: The starting dose will be 300 mg niraparib (or modified according to patient weight and platelet count), taken orally once a day for each cycle of 28 days.
Period: Overall Study
Arm/Group | Niraparib Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Niraparib Treatment: Patients were treated with individualized starting dose of Niraparib.
  Niraparib: The starting dose was 300 mg niraparib (or modified according to patient weight and platelet count), taken orally once a day for each cycle of 28 days.
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9
Primary Site of Cancer [Number; unit: number of participants]
  Astrocytoma | 2
  GBM | 6
  Oligodendroglioma | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience Adverse Events
Description: Number of patients who experience adverse events with individualized starting dose (ISD) of niraparib using CTCAE v5.0
Time Frame: Up to 17 months
Population: All patients enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Efficacy of Treatment in Dose Expansion Phase
Description: Percentage of patients who respond to niraparib monitored by disease control rate (stable disease and better) using RANO from start of treatment for up to 12 months.
Time Frame: up to 12 months
Population: study terminated early, only 6 participants in dose expansion phase.
Measure: Number; unit: participants
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 6
participants | 0

3. Primary Outcome: Number of Patients Who Experience Toxicities With Individualized Starting Dose (ISD) of Niraparib Using CTCAE v5.0
Description: Number of patients who experience toxicities (defined as grade 3 or 4 adverse events) with individualized starting dose (ISD) of niraparib using CTCAE v5.0
Time Frame: 5 months
Population: Patients who received at least one dose of Niraparib
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 9
Participants | 5

4. Secondary Outcome: Progression Free Survival in Dose Expansion Phase
Description: Proportion of patients who have progression-free survival from date of study entry until the first documented date of progression or date of death, whichever comes first.
Time Frame: 20 months
Population: Patients who enrolled in study and took at least one dose of study drug. Patient must be in the dose expansion phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 6
Months | 1.62 [1.06 to NA] — The upper bound confidence interval never dropped before the 50% margin and therefore cannot be calculated.

5. Secondary Outcome: Overall Survival in Dose Expansion Phase
Description: Proportion of patients with overall survival on the study defined as time from date of study entry to death by any cause.
Time Frame: 20 months
Population: Patients who enrolled in study and consumed at least one dose of study drug. Patient must be in the dose expansion phase
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 6
Months | 10.81 [4.63 to NA] — The upper bound confidence interval never passed the 50% margin and therefore cannot be calculated.

6. Secondary Outcome: Duration of Disease Control of All Patients
Description: Duration of response in patients treated with niraparib defined as time from date of first response (stable disease or better) to the first date of non-response post treatment on the study.
Time Frame: up to 4 years
Population: Outcome measure was not calculated due to early study termination-- no patients experienced response to treatment. Due to this, we cannot calculate a duration of response because we don't have any responders to evaluate
Arm/Group | Niraparib Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 17 months.
Description: CTCAE 5.0
Groups:
- Niraparib Treatment: Patients will be treated with individualized starting dose of Niraparib. Since each patient's dose will be individualized based on patients' weight and platelet count, arms/groups are combined.
  Niraparib: The starting dose will be 300 mg niraparib (or modified according to patient weight and platelet count), taken orally once a day for each cycle of 28 days.
Arm/Group | Niraparib Treatment
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib Treatment (N=9)
Death NOS (General disorders) | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib Treatment (N=9)
Anemia (Blood and lymphatic system disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 6
Gait disturbance (General disorders) | 2
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Hemoglobin increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 5
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT05297864/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05297864/SAP_001.pdf